CLINICAL TRIAL: NCT05182853
Title: Voiding Disorders in Children After Sacrococcygeal Teratoma Resection
Acronym: TSC-URO
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0377
Record Dates: First submitted 2021-12-22; First posted 2022-01-10 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Sacrococcygeal Teratoma; Neurogenic Bladder; Voiding Disorders
Keywords: Teratoma; sacrococcygeal region; urinary incontinence; neurogenic bladder; children
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Teratoma; Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sacrococcygeal teratomas are the most common neonatal tumors and require rapid and complete resection. Tumor nerve compression and pelvic surgical sequelae may lead to many and varied voiding disorders. Data concerning long-term vesico-sphincteric disorders are conflicting. Some studies find good functional results [Cozzi et al., 2008; Draper et al., 2009]. However other authors reveal neurologic bladder with detrusor sphincter dyssynergia [Hambraeus et al., 2018] and rise concerned about long-term renal function [Khanna et al., 2019; Rehfuss et al., 2020] even in the absence of clinical voiding disorders. Most of studies include young patients with other malformations such as anorectal malformations or dysraphisms which may impact the results. The main objective is to assess bladder dysfunction in children aged 6 to 18 years after isolated sacrococcygeal teratoma resection.

ELIGIBILITY:
Inclusion criteria:

* Children aged 6 to 18
* history of sacrococcygeal teratoma resection

Exclusion criteria:

* Associated anorectal malformation
* Associated neurological pathology

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who underwent surgical treatment of a sacrococcygeal teratoma, without ano rectal malformation or any other neurological pathology
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Presence of voiding disorders | Day 1
  Presence of voiding disorders will be assessed by the scale: Dysfonctional voiding scoring system

SECONDARY OUTCOMES:
Presence of defecation disorders | Day 1
  The Presence of defecation disorders will be assessed by the scale: Bristol stool scale
Presence of secondary neurological bladder | Day 1
  the Presence of secondary neurological bladder will be assessed by the uroflowmetry

CONTACTS AND LOCATIONS:
Overall Officials: Sarah GARNIER, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC